CLINICAL TRIAL: NCT02235675
Title: Prospective, Multicenter Tack Optimized Balloon Angioplasty Below the Knee (TOBA - BTK) Study for Infrapopliteal Arteries Using the Tack-It Endovascular System™
Brief Title: Tack Optimized Balloon Angioplasty Below the Knee (TOBA - BTK) Study
Acronym: TOBABTK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TD 0109
Record Dates: First submitted 2014-09-04; First posted 2014-09-10 (Estimated); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Critical Limb Ischemia; Peripheral Artery Disease
Keywords: Angioplasty; Peripheral Artery Disease; Critical Limb Ischemia; CLI; PAD
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tack-It (Experimental): Implant of the Intact Vascular Tack-It Endovascular System to repair post angioplasty dissections.
  Interventions: Device: Tack-It Endovascular System

INTERVENTIONS:
Device: Tack-It Endovascular System — Repair of post-PTA dissections using the Intact Vascular Tack-It implant.
  Other Names: Tack-It Dissection Repair; Intact Vascular Tack-It; Tack-It; Tack

SUMMARY:
Multi-center study to optimize below the knee (BTK) balloon angioplasty results by creating tissue apposition in peripheral arteries with Reference Vessel Diameter's (RVD) ranging from 1.5mm to 4.5mm.

DETAILED DESCRIPTION:
This first in man (FIM) study is to collect data in support of the safety and performance of the Intact Vascular Tack-It Endovascular System™ for tissue apposition to optimize balloon angioplasty.

Study primary endpoints:

Safety: Composite of Major Adverse Limb Events (MALE) and Peri-procedural Death (POD), assessed at 1 month. Endpoint includes any of the following:

* Major amputation - amputation above the ankle
* Re-intervention (surgical or endovascular) in the target limb
* Procedure-related death - any death within 1 month of the index procedure or any MALE

Device Success: The achievement of successful delivery and deployment of the study device(s) at the intended target site(s) and successful withdrawal of the delivery catheter.

Technical Success: Device success (defined above) and the ability of the Tack to resolve post-PTA dissection, demonstrating angiographic patency at the conclusion of the procedure.

Clinical Success: Ability of the Tack to resolve post-PTA dissection and achieve patency at the conclusion of the procedure, without procedure related complications within 48 hours after the index procedure or at hospital discharge, whichever is sooner.

Study secondary endpoints:

The following events will be assessed at 3, 6 and 12 months:

* All-cause mortality
* Amputation of the limb (above the ankle)
* Amputation free survival
* Clinically driven target vessel revascularization (TVR)
* Clinically driven target lesion revascularization (TLR)
* Changes in Rutherford Clinical Category from baseline

The following parameters will be assessed at 1, 3, 6 and 12 months:

* Maintenance of luminal patency of the target lesion by TBI (≤0.15 decrease) as compared to the baseline TBI obtained prior to discharge
* Doppler Exam (presence of signal)

Study observational endpoint:

The following parameter will be assessed at 6 months (Per local Standard of Care):

• Angiographic percent diameter stenosis

ELIGIBILITY:
Inclusion Criteria:

* Age of subject is >18
* Subject or subject's legal representative has been informed of the nature of the study, agrees to participate and has signed the consent form
* Subject has critical limb ischemia (CLI)
* Subject has Rutherford Clinical Category 4-5. (hemodynamic reference)
* Reference vessel diameter below the knee (BTK) is between 1.5mm and 4.5mm (inclusive).
* De-novo target lesion(s) has stenosis >70%.
* Must be able to perform PTA. The PTA must result in a dissection Type A - F at some location along the treatment site.
* Any vessel intervened on must have distal reconstitution above the ankle.
* Inflow Iliac, SFA and Popliteal lesions can be treated during the same procedure using standard angioplasty and/or an approved device. These inflow lesions must be treated first, prior to consideration of treatment of BTK lesions. The patient can be enrolled if the inflow lesions are treated with good angiographic results (must have <30% residual stenosis and no evidence of embolization).

Key Exclusion Criteria:

* The subject has a lesion on the plantar surface of the heel or over the Achilles tendon or has exposed calcaneus.
* The subject has extensive forefoot gangrene / ischemic ulcer that cannot be resolved with standard metatarsal amputation.
* Previous treatment failure of inflow arteries (Iliac, SFA and Popliteal)
* Subject with below knee bypass.
* Subject has significant stenosis or occlusion of inflow vessels tract (proximal disease) not successfully treated (>30% residual stenosis and/or complication of the procedure) prior to BTK angioplasty and patient enrollment.
* Subject is permanently wheel-chair bound or bedridden.
* Subject has an allergy to contrast medium that cannot be pretreated.
* Episode of acute limb ischemia within the previous 30 days.
* Subject is undergoing atherectomy in the target limb or cryoplasty or stenting of BTK treatment site.
* Subject has a systemic infection with positive blood cultures/bacteremia within one week.
* Subject has undrained pus or spreading wet gangrene in the foot that is not controlled at the time of revascularization procedure.
* Subject in whom antiplatelet, anticoagulant, or thrombolytic therapy is contraindicated.
* Myocardial infarction within 30 days prior to enrollment.
* History of stroke within 180 days prior to enrollment.
* Subject has acute or chronic renal disease (e.g., as measured by a serum creatinine of >2.5 mg/dL or >220 umol/L).
* Subject has a known hypersensitivity or contraindication to nitinol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-12; Primary Completion 2016-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Primary Endpoints | 30 Days
  Safety: Composite of Major Adverse Limb Events (MALE) and Peri-procedural Death (POD), assessed at 1 month. Endpoint includes any of the following:
  * Major amputation - amputation above the ankle
  * Re-intervention (surgical or endovascular) in the target limb
  * Procedure-related death - any death within 1 month of the index procedure or any MALE

SECONDARY OUTCOMES:
Secondary Endpoints | 1, 3, 6 and 12 Months
  The composite of following events will be assessed at 3, 6 and 12 months or as noted:
  * All-cause mortality
  * Amputation of the limb (above the ankle)
  * Amputation free survival
  * Clinically driven target vessel revascularization (TVR)
  * Clinically driven target lesion revascularization (TLR)
  * Changes in Rutherford Clinical Category from baseline
  * Maintenance of luminal patency of the target lesion by TBI (≤0.15 decrease) as compared to the baseline TBI obtained prior to discharge at 1,3,6 and 12 months.
  * Doppler Exam (presence of signal at 1,3,6 and 12 months)

OTHER OUTCOMES:
Observational Endpoint | 6 Months
  The following parameter will be assessed at 6 months (Per local Standard of Care):
  • Angiographic percent diameter stenosis

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Brodmann, MD, Principal Investigator — MEDIZINISCHE UNIVERSITAT GRAZ
Locations (1):
- Medizinische Universitat Graz, Graz, Austria